CLINICAL TRIAL: NCT05585190
Title: Stand Up for Your Health: a Randomized Study
Brief Title: Stand Up for Your Health with a Sit-stand Desk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jacquelyn Kulinski, Principal Investigator, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 44431
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pre Diabetes; Obesity; Metabolic Syndrome; Sedentary Behavior
Keywords: Pre Diabetes; Obesity; Metabolic Syndrome; Cardiovascular; Sit-stand desk; Physical Activity; Overweight; Sedentary; Standing desk; Insulin resistance
MeSH Terms: conditions — Glucose Intolerance; Obesity; Metabolic Syndrome; Sedentary Behavior; Motor Activity; Overweight; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Other): Subjects will not receive a sit/stand desk for the duration of the study and will be asked to follow their normal work day routine.
  Interventions: Other: Control
- 2-Hour Group (Active Comparator): Sit-stand desk intervention group, subjects are asked to maintain the desk in the standing position at LEAST 2 hours each work day.
  Interventions: Other: Sit-Stand Desk at Work
- 3-Hour Group (Active Comparator): Sit-stand desk intervention group, subjects are asked to maintain the desk in the standing position at LEAST 3 hours each work day.
  Interventions: Other: Sit-Stand Desk at Work

INTERVENTIONS:
Other: Control — No intervention.
  Arms: Control
Other: Sit-Stand Desk at Work — Subjects will receive a sit-stand desk at their work location.
  Arms: 2-Hour Group; 3-Hour Group

SUMMARY:
More than 84 million - or 1 out of every 3 U.S. adults - have prediabetes, a condition that if not treated often leads to type 2 diabetes within five years. Average medical expenditures among diabetics are about 2.3 times higher than expenditures for people without diabetes. Physical inactivity and elevated body mass index (BMI) are major risk factors for the disease. Sedentary behavior is becoming increasingly prevalent with the growth of a 'work from home' culture, most recently driven by the COVID-19 pandemic. Cross-sectional epidemiologic data report significant associations between high amounts of sedentary (sitting) time and prevalent cardiovascular disease and diabetes. In our pilot study of 15 subjects with sedentary office jobs, 6 months of sit-stand desk use resulted in a 23% improvement in insulin resistance, most substantial in those who decreased daily sitting by over 90 minutes/day. Additional improvements in vascular endothelial function and triglyceride levels were seen without any change in exercise activity, step counts, or body weight. These findings not only corroborate epidemiologic findings on this topic but suggest causality and warrant a randomized control trial.

The investigators hypothesize that adult subjects at-risk for diabetes will improve insulin sensitivity, metabolic and vascular (endothelial) health with a sit-stand desk intervention at work (whether in the office or at home), in the context of a randomized, controlled trial. The investigators will randomize 198 sedentary office workers with a BMI≥25 at risk for type 2 diabetes mellitus in a 1:1:1 ratio of three groups: (a) sit-stand desk intervention targeting 2 hours standing per day; (b) sit-stand desk intervention targeting 3 hours standing per day; or (c) control arm over 6 months. The block randomization design will allow for important dose-response analyses.

The investigators will objectively quantify standing time, sedentary time, sedentary bouts, daily steps, and exercise activity times using a compact and re-usable accelerometer that adheres to the subject's thigh. This will provide objective assessments of activity levels and sedentary times for 7 full days each at baseline, 3 and 6 months. The device is equipped with an inclinometer to classify posture (sitting verses standing).

ELIGIBILITY:
Inclusion Criteria:

1. Overweight or obese (body mass index of 25 kg/m2 or higher)
2. Employees with "sedentary" jobs, defined as spending at least 75% of their (8 hours or more) workday sitting at a desk (at home or in an office)
3. Defined as "at-risk" for diabetes, defined as either:

   1. Prediabetes (HbA1c of 5.7% to 6.4%) or a fasting glucose of 100 to 125 mg/dL
   2. Having one or more additional risk factors: (beyond BMI>25)

      * Age 45 years or older
      * Family history of diabetes mellitus in a first-degree relative
      * Physical inactivity (no structured exercise activity)
      * History of gestational diabetes, hypertension, or dyslipidemia
      * African American, Alaska Native, American Indian, Asian American, Hispanic/Latino, Native Hawaiian, or Pacific Islander ethnicity

Exclusion Criteria:

1. Established cardiovascular disease (myocardial infarction, coronary stent, coronary artery bypass grafting, cardiac transplant, or angina)
2. Established congestive heart failure or cardiomyopathy
3. Established peripheral vascular disease
4. Established diabetes (HbA1c ≥ 6.5% or on diabetes medications or insulin)
5. Chronic musculoskeletal disorders involving the lower extremities, such as arthritis of the knees or hips, or regular use of ambulatory assist devices such as a walker or cane
6. Neuropathy of any etiology
7. Positional syncope or history of orthostasis
8. Less than 4 days/week at any single office (or work-from-home) location.
9. Current use of a standing desk for work
10. Tobacco use within the previous 12 months
11. Current illicit drug use or excessive alcohol use (defined as more than 14 drinks/week for women, more than 28 drinks/week for men)
12. Steroid use ≥21 days/year
13. Fasting triglyceride level ≥ 500 mg/dL
14. Thyroid disease
15. Uncontrolled or untreated hypertension(>150/90 mm Hg)
16. Pregnant or lactating (or plans to become pregnant in the next 6 months)
17. LDL cholesterol ≥ 190mg/dL
18. Currently enrolled or plans to diet or join a weight loss program over the next 6 months.
19. Non-English speaker

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity (HOMA-IR) | change from baseline to 6 months
  Determine if use of a sit-stand desk improves insulin sensitivity and ascertain if there is a dose-response relationship with changes in sedentary time.

SECONDARY OUTCOMES:
HbA1c | change from baseline to 6 months
  Determine if use of a sit-stand desk improves HbA1c.
fasting glucose | change from baseline to 6 months
  Determine if use of a sit-stand desk improves fasting glucose.
fasting insulin level | change from baseline to 6 months
  Determine if use of a sit-stand desk improves (reduces) fasting insulin levels.
metabolic syndrome severity (MetS) score | change from baseline to 6 months
  Determine if use of a sit-stand desk at work improves metabolic health, as assessed by the MetS severity score, in sedentary office workers at-risk for type 2 diabetes mellitus.
metabolic syndrome | change from baseline to 6 months
  Determine if use of a sit-stand desk at work improves metabolic health, as assessed by number of (NCEP ATP III) metabolic syndrome criteria, in sedentary office workers at-risk for type 2 diabetes mellitus.
fasting triglycerides | change from baseline to 6 months
  To quantify changes in serum fasting triglyceride levels with the sit-stand desk (compared to no desk), while accounting for dietary intake.
very low-density lipoprotein (VLDL) particle number | change from baseline to 6 months
  To quantify changes in serum triglyceride-rich, remnant lipoproteins with the sit-stand desk (compared to no desk), while accounting for dietary intake.
vascular endothelial function (superficial femoral artery) | change from baseline to 6 months
  To measure the changes in vascular endothelial function with the sit-stand desk compared to control.

OTHER OUTCOMES:
Acceptability Questionnaire | 6 months
  Includes questions on ease of use, comfort, perceived work productivity, and musculoskeletal discomforts related to use of the sit-stand desk. Higher scores are more favorable.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Within 1 year of completion of all studies procedures

REFERENCES:
- [Background] Bodker A, Visotcky A, Gutterman D, Widlansky ME, Kulinski J. The impact of standing desks on cardiometabolic and vascular health. Vasc Med. 2021 Aug;26(4):374-382. doi: 10.1177/1358863X211001934. Epub 2021 Apr 5. PMID 33813968
- [Derived] Hammad M, Shankar S, Gao Y, Kulinski J. Stand up for your health: Rationale and design for a randomized controlled trial. Contemp Clin Trials. 2026 Feb;161:108216. doi: 10.1016/j.cct.2026.108216. Epub 2026 Jan 6. PMID 41506470